CLINICAL TRIAL: NCT06436352
Title: Does Capsulotomy in Closed Reduction of Femoral Neck Fractures Decrease Incidence of Avascular Necrosis?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Omar Sabry, Dr., Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-143-2019
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: A prospective research was carried out between January 2021 and February 2023. Patients were randomized into two groups: Group I: cases with capsulotomy and Group II: cases without capsulotomy. The study was conducted after an ethical approval was obtained.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: cases with capsulotomy during fixation (Experimental): before fixation, We perform a guide wire insertion passing anterior to the Greater Trochanter and the neck is done. then passing a pointed Schanz 5 or 6mm ± scalpel, under X-ray in AP-lateral views until reaching the capsule (intra trochanteric line). Aspiration of hematoma with suction was done.
  Interventions: Procedure: Capsulotomy and fixation
- Group II: cases without capsulotomy during fixation (Active Comparator): we fix the fracture without capsulotomy
  Interventions: Procedure: Fixation only

INTERVENTIONS:
Procedure: Capsulotomy and fixation — Firstly, Guide wire insertion passing anterior to the GT and the neck is done. then passing a pointed Schanze 5 or 6 ± scalpel, under X-ray in AP-lateral views until reaching the capsule (intra trochanteric line). Aspiration of hematoma with suction was done.
  Then we fix the fracture by proceeding with drilling over the wires using a "3.6 mm cannulated drill bit". Then, we place three "7.0 mm or 7.3 mm cannulated cancellous screws" over the wires. In younger patients with thick cancellous bone, a "cannulated tap" may be required to precut the thread. A washer may be used to prevent the screw head from penetrating the thin cortex.
  Arms: Group I: cases with capsulotomy during fixation
Procedure: Fixation only — we fix the fracture by proceeding with drilling over the wires using a "3.6 mm cannulated drill bit". Then, we place three "7.0 mm or 7.3 mm cannulated cancellous screws" over the wires. In younger patients with thick cancellous bone, a "cannulated tap" may be required to precut the thread. A washer may be used to prevent the screw head from penetrating the thin cortex.
  Arms: Group II: cases without capsulotomy during fixation

SUMMARY:
Femur's neck injuries are frequently encountered fractures. They are usually due to high energy or low energy indirect trauma. Healing of these fractures is usually hindered due to "avascular necrosis (AVN)" or "non-union" of the Femur's head. This study looks forward to investigating the impact of capsulotomy and internal fixation in lowering the incidence of complications and improving the functional outcomes.

DETAILED DESCRIPTION:
Femoral neck fractures constitute a frequent orthopaedic, usually due to indirect assault. It primarily affects older people, with younger people accounting for barely 2 - 3%. Nevertheless, since transportation has recently advanced rapidly, high-energy trauma has become increasingly widespread. The prevalence of femur neck injuries among youth is likewise growing in hospitals by an estimated rate of about 6000 yearly. Hip blood supply is especially important while addressing femoral neck fractures. Blood supply emerges from the capsular, intramedullary, and the ligamentum teres vessels. In adults, capsular vessels provide most of the femur's head blood supply. The arteries originate out of the "medial and lateral circumflex femoral arteries". Those areteries are in turn branced out of the profunda femoris in seventy nine of the population. There is an exception for 20% of population where one vessel originates from the femoral artery. Moreover, there is 1% of the population in which both vessels originate from the femoral artery. The effectiveness and benefits of capsulotomy in treating femur's neck fractures among youth were compared to "closed reduction and internal fixation (CRIF)". AVN and non-union are the most prevalent and difficult complications. In terms of "trauma degree index" (incision length, amount of lost blood, and operative time), capsulotomy and internal fixation are less effective than CRIF. However, it outperforms CRIF in functional effectiveness (Harris Hip Score.

Some differences exist between capsulotomy reduction and internal fixation. First and foremost is proper anatomical reduction. With direct sight and adequate exposure, an acceptable anatomical reduction can be obtained, laying the groundwork for the healing of fractures. Furthermore, it could unlock certain retinacular arteries that have been temporarily blocked by kinking or stretching, allowing for the the restoration of some vascular function. The second principal is "stable internal fixation" that can be achieved by proper placement of the screws under direct visualization.

Researchers have concluded that evacuating of the hematoma significantly lowers the capsular pressure and improves pulse perfusion of the femur's head. Our study aims to investigate the efficiency of capsulotomy in enhancing the healing process of femur's neck fractures.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature patients with fracture neck femur who will undergo urgent surgery within 48 hours.
* Male and female patients of any garden classification of femoral neck fractures
* within age group from 18 - 55 years

Exclusion Criteria:

* Patients of age below 18 years or above 55 years.
* those with metabolic bone disease, pathological fractures, stress fracture or delayed presentation more than 48 hours were excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Harris hip score | 6 months
  The HHS is a measure of dysfunction so the higher the score, the better the outcome for the individual. Results can be recorded and calculated online. The maximum score possible is 100. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.

SECONDARY OUTCOMES:
Intra-operative blood loss | during the operation
  in ml

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy Hospital - Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No